CLINICAL TRIAL: NCT02563002
Title: A Phase III Study of Pembrolizumab (MK-3475) vs. Chemotherapy in Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Stage IV Colorectal Carcinoma (KEYNOTE-177)
Brief Title: Study of Pembrolizumab (MK-3475) vs Standard Therapy in Participants With Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) Stage IV Colorectal Carcinoma (MK-3475-177/KEYNOTE-177)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-177; 163238 (Registry Identifier: JAPIC-CTI); MK-3475-177 (Other: MSD); KEYNOTE-177 (Other: MSD); 2015-002024-89 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2022-03-16 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Carcinoma
Keywords: Programmed Cell Death Receptor 1 (PD-1); Programmed Cell Death Receptor Ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Colorectal Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — IFL protocol; pembrolizumab; Bevacizumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 treatments (approximately 2 years). Participants that have stopped the initial course of pembrolizumab and have stable disease but progress after discontinuation can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 year additional).
  Interventions: Biological: Pembrolizumab
- Standard of Care (SOC) (Active Comparator): Participants receive 1 of 6 possible standard chemotherapy regimens: mFOLFOX6, or mFOLFOX6+bevacizumab 5 mg/kg IV on Day 1 of each 2-week cycle, or mFOLFOX6+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly in each 2-week cycle, or FOLFIRI, or FOLFIRI+bevacizumab 5 mg/kg IV on Day 1 of each 2-week cycle, or FOLFIRI+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly in each 2-week cycle. Participants with documented disease progression following chemotherapy can crossover to receive pembrolizumab for up to 35 cycles (approximately 2 years). Participants that have stopped pembrolizumab and have stable disease but progress after discontinuation can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 year additional).
  Interventions: Drug: mFOLFOX6; Drug: FOLFIRI; Biological: Pembrolizumab; Biological: Bevacizumab; Biological: Cetuximab

INTERVENTIONS:
Drug: mFOLFOX6 — Regimen consists of oxaliplatin 85 mg/m^2 IV on Day 1, leucovorin 400 mg/m^2 or levoleucovorin 200 mg/m^2 IV on Day 1, 5-fluorouracil (5-FU) 400 mg/m^2 IV bolus on Day 1 and then 1200 mg/m^2/day IV over 2 days for total dose of 2400 mg/m^2 in each 2-week cycle
  Arms: Standard of Care (SOC)
Drug: FOLFIRI — Regimen consists of irinotecan 180 mg/m^2 IV on Day 1, leucovorin 400 mg/m^2 or levoleucovorin 200 mg/m^2 IV on Day 1, 5-FU 400 mg/m^2 IV bolus on Day 1 and then 1200 mg/m^2/day IV over 2 days for total dose of 2400 mg/m^2 in each 2-week cycle
  Arms: Standard of Care (SOC)
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; SCH 900475; KEYTRUDA®
Biological: Bevacizumab — IV infusion
  Arms: Standard of Care (SOC)
Biological: Cetuximab — IV infusion
  Arms: Standard of Care (SOC)

SUMMARY:
In this study, participants with stage IV Microsatellite Instability-High (MSI-H) or Mismatch Repair Deficient (dMMR) colorectal carcinoma (CRC) will be randomly assigned to receive either pembrolizumab or the Investigator's choice of 1 of 6 standard of care (SOC) chemotherapy regimens for the treatment of advanced colorectal carcinoma. The primary study hypothesis is that pembrolizumab will prolong progression-free survival (PFS) or overall survival (OS) compared to current SOC chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally confirmed dMMR or MSI-H stage IV colorectal carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days prior to study start
* Life expectancy of at least 3 months
* Measurable disease
* Female participants of childbearing potential must be willing to use adequate contraception for the course of the study starting with the first dose of study medication through 180 days after the last dose of standard of care (SOC) therapy or 120 days after the last pembrolizumab dose
* Male participants must agree to use adequate contraception for the course of the study starting with the first dose of study medication through 180 days after the last dose of study medication for chemotherapy arm (no contraception requirement for pembrolizumab [MK-3475] arm)
* Adequate organ function

Exclusion Criteria:

* Has received prior systemic therapy for Stage IV colorectal cancer. May have received prior adjuvant chemotherapy for colorectal cancer as long as it was completed at least 6 months prior to randomization on this study
* Currently participating and receiving treatment in another study, or participated in a study of an investigational agent and received treatment, or used an investigational device within 4 weeks of randomization
* Active autoimmune disease that has required systemic treatment in past 2 years
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization on this study
* Radiation therapy within 4 weeks prior to randomization on this study and not recovered to baseline from adverse events due to radiation therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomization on this study
* Has received prior therapy with an immune checkpoint inhibitor (e.g., anti-programmed cell death [PD]-1, anti-PD ligand 1 [L1], anti-PD-L2 agent, or anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4] agent, etc.)
* Another malignancy that is progressing or requires active treatment with the exception of non-melanomatous skin cancer that has undergone potentially curative therapy and in situ cervical carcinoma
* Received a live or a live attenuated vaccine within 30 days of planned start of study medication
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B or C
* Known history of, or any evidence of interstitial lung disease or active, non-infectious pneumonitis
* Known history of active tuberculosis (Bacillus tuberculosis [TB])
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of SOC (for male and female participants) or 120 days after the last dose of pembrolizumab (for female participants only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Yoshino T, Andre T, Kim TW, Yong WP, Shiu KK, Jensen BV, Jensen LH, Punt CJA, Smith D, Garcia-Carbonero R, Alcaide-Garcia J, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Le DT, Adachi N, Fogelman D, Marinello P, Diaz LA Jr. Pembrolizumab in Asian patients with microsatellite-instability-high/mismatch-repair-deficient colorectal cancer. Cancer Sci. 2023 Mar;114(3):1026-1036. doi: 10.1111/cas.15650. Epub 2022 Dec 12. PMID 36369901
- [Derived] Diaz LA Jr, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fourchardiere C, Rivera F, Elez E, Le DT, Yoshino T, Zhong WY, Fogelman D, Marinello P, Andre T; KEYNOTE-177 Investigators. Pembrolizumab versus chemotherapy for microsatellite instability-high or mismatch repair-deficient metastatic colorectal cancer (KEYNOTE-177): final analysis of a randomised, open-label, phase 3 study. Lancet Oncol. 2022 May;23(5):659-670. doi: 10.1016/S1470-2045(22)00197-8. Epub 2022 Apr 12. PMID 35427471
- [Derived] Andre T, Amonkar M, Norquist JM, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt CJA, Smith D, Garcia-Carbonero R, Sevilla I, De La Fouchardiere C, Rivera F, Elez E, Diaz LA Jr, Yoshino T, Van Cutsem E, Yang P, Farooqui M, Le DT. Health-related quality of life in patients with microsatellite instability-high or mismatch repair deficient metastatic colorectal cancer treated with first-line pembrolizumab versus chemotherapy (KEYNOTE-177): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 May;22(5):665-677. doi: 10.1016/S1470-2045(21)00064-4. Epub 2021 Apr 1. PMID 33812497
- [Derived] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26099&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 307 participants randomized in the study, 296 participants received study medication and were evaluable for safety analyses.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 treatments (approximately 2 years). Eligible participants who stopped the initial course of pembrolizumab due to complete response (CR) or completed initial course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
- Standard of Care (SOC): Participants received 1 of 6 possible standard chemotherapy regimens: mFOLFOX6, or mFOLFOX6+bevacizumab 5 mg/kg IV on Day 1 of each 2-week cycle, or mFOLFOX6+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly in each 2-week cycle, or FOLFIRI, or FOLFIRI+bevacizumab 5 mg/kg IV on Day 1 of each 2-week cycle, or FOLFIRI+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly in each 2-week cycle. Participants with documented disease progression following chemotherapy can crossover to receive pembrolizumab for up to 35 cycles (approximately 2 years). Eligible cross over participants who stopped pembrolizumab who stopped pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
Period: Overall Study
Arm/Group | Pembrolizumab | Standard of Care (SOC)
Started | 153 | 154
Treated | 153 | 143
Received Second Course of Pembrolizumab | 12 | 5
Switched Over to Pembrolizumab | 0 | 7
Completed | 0 | 0
Not Completed | 153 | 154
Not completed — Death | 72 | 87
Not completed — Lost to Follow-up | 5 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 2 | 10
Not completed — Sponsor decision | 74 | 55

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Standard of Care (SOC) | Total
Number analyzed (Participants) | 153 | 154 | 307
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (14.9) | 60.6 (14.8) | 61.2 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 72 | 154
  Male | 71 | 82 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 128 | 131 | 259
  Unknown or Not Reported | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 26 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 5 | 14
  White | 113 | 116 | 229
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per RECIST1.1 As Assessed by Central Imaging Vendor
Description: PFS was defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 based on blinded central imaging vendor review or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. Hazards ratio (HR) and associated 95% confidence intervals (CIs) from a Cox proportional hazard model with Efron's method of tie handling and with a single treatment covariate was presented for the first course study treatment per protocol.
Time Frame: Up to approximately 59 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard of Care (SOC)
Number analyzed (Participants) | 153 | 154
Months | 16.5 [5.4 to 38.1] | 8.2 [6.1 to 10.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard of Care (SOC); Test type: Other; p = 0.0001, Log Rank; One-sided p-value based on log rank test; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.45 to 0.79] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of analysis were censored at the date of last known contact. HR and associated 95% CIs from a Cox proportional hazard model with Efron's method of tie handling and with a single treatment covariate was presented for the first course study treatment per protocol.
Time Frame: Up to approximately 59 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard of Care (SOC)
Number analyzed (Participants) | 153 | 154
Months | NA [49.2 to NA] — Median OS and upper limit for OS was not reached at the time of last disease assessment due to insufficient number of participants with events. | 36.7 [27.6 to NA] — Upper limit for OS was not reached at the time of last disease assessment due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard of Care (SOC); Test type: Other; p = 0.0359, Log Rank; One-sided p-value based on log rank test; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.53 to 1.03] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate

3. Secondary Outcome: Overall Response Rate (ORR) Per RECIST1.1 as Assessed by Central Imaging Vendor
Description: ORR was defined as the percentage of the participants who experienced a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 as assessed by the central imaging vendor. The percentage of participants who experienced a CR or PR was presented for the first course of study treatment per protocol.
Time Frame: Up to approximately 59 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard of Care (SOC)
Number analyzed (Participants) | 153 | 154
Percentage of Participants | 45.1 [37.1 to 53.3] | 33.1 [25.8 to 41.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard of Care (SOC); Test type: Other; p = 0.0159, Miettinen & Nurminen method — One-sided p-value based on Miettinen & Nurminen method; Difference in percentage = 12.0, 95% CI 2-sided [1.0 to 22.6] — Based on Miettinen & Nurminen method

4. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE was presented for the first course study treatment per protocol.
Time Frame: Up to approximately 59 months
Population: All participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Standard of Care (SOC)
Number analyzed (Participants) | 153 | 143
Participants | 149 | 142

5. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change infrequency and/or intensity) of a preexisting condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE was presented for the first course study treatment per protocol.
Time Frame: Up to approximately 59 months
Population: All participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Standard of Care (SOC)
Number analyzed (Participants) | 153 | 143
Participants | 21 | 20

ADVERSE EVENTS:
Time Frame: Up to approximately 91 months
Description: All-cause mortality (ACM)=all randomized participants. AEs=all participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression (NP), malignant NP, and disease progression not related to treatment are excluded. Per protocol, collection of AEs and ACM were planned to be done in first and second courses.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 treatments (approximately 2 years).
- Standard of Care (SOC) First Course: Participants received 1 of 6 possible standard chemotherapy regimens: mFOLFOX6, or mFOLFOX6+bevacizumab 5 mg/kg IV on Day 1 of each 2-week cycle, or mFOLFOX6+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly in each 2-week cycle, or FOLFIRI, or FOLFIRI+bevacizumab 5 mg/kg IV on Day 1 of each 2-week cycle, or FOLFIRI+cetuximab 400 mg/m^2 IV over 2 hours then 250 mg/m^2 over 1 hour weekly in each 2-week cycle.
- SOC Switched Over to Pembrolizumab: Eligible participants with documented disease progression following chemotherapy in SOC arm switched over to receive pembrolizumab for up to 35 cycles (approximately 2 years).
- Pembrolizumab Second Course: Participants who received pembrolizumab as a first course and stopped the first course of pembrolizumab due to complete response (CR) or completed the first course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
- SOC Switched Over to Pembrolizumab-Second Course: Participants who switched over from SOC and received pembrolizumab and subsequently stopped the first course of pembrolizumab due to complete response (CR) or completed the first course of pembrolizumab and had stable disease but progressed after discontinuation, initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (approximately 1 year additional).
Arm/Group | Pembrolizumab First Course | Standard of Care (SOC) First Course | SOC Switched Over to Pembrolizumab | Pembrolizumab Second Course | SOC Switched Over to Pembrolizumab-Second Course
All-Cause Mortality (participants affected / at risk) | 68/153 | 58/154 | 30/57 | 4/12 | 2/5
Serious Adverse Events (participants affected / at risk) | 62/153 | 76/143 | 27/57 | 3/12 | 1/5
Other Adverse Events (participants affected / at risk) | 145/153 | 142/143 | 53/57 | 11/12 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=153) | Standard of Care (SOC) First Course (N=143) | SOC Switched Over to Pembrolizumab (N=57) | Pembrolizumab Second Course (N=12) | SOC Switched Over to Pembrolizumab-Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 9 (9) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 5 (9) | 3 (3) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningoencephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stoma site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Norovirus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudobulbar palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Autoimmune nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=153) | Standard of Care (SOC) First Course (N=143) | SOC Switched Over to Pembrolizumab (N=57) | Pembrolizumab Second Course (N=12) | SOC Switched Over to Pembrolizumab-Second Course (N=5)
Anaemia (Blood and lymphatic system disorders) | 26 (32) | 33 (40) | 9 (18) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (12) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 27 (52) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 8 (18) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 6 (6) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 19 (20) | 4 (6) | 7 (7) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 9 (11) | 3 (4) | 0 (0) | 1 (2) | 0 (0)
Ocular hyperaemia (Eye disorders) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 8 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 34 (56) | 41 (62) | 8 (12) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 19 (21) | 11 (14) | 2 (3) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 26 (30) | 45 (76) | 13 (19) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 65 (107) | 89 (204) | 17 (36) | 2 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 17 (18) | 9 (10) | 4 (5) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 16 (21) | 5 (7) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 6 (8) | 1 (1) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 47 (69) | 85 (283) | 16 (23) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 10 (11) | 43 (75) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 33 (53) | 53 (85) | 12 (20) | 0 (0) | 0 (0)
Asthenia (General disorders) | 19 (32) | 30 (57) | 5 (8) | 1 (1) | 0 (0)
Chest pain (General disorders) | 8 (9) | 3 (4) | 4 (5) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (5) | 7 (9) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 58 (79) | 70 (176) | 9 (9) | 2 (3) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 14 (20) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Malaise (General disorders) | 10 (11) | 6 (8) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 7 (7) | 27 (49) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 18 (24) | 11 (13) | 10 (11) | 0 (0) | 0 (0)
Pain (General disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 4 (5) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 24 (29) | 20 (28) | 7 (9) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 1 (2) | 8 (12) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 4 (4) | 5 (8) | 4 (6) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 7 (8) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (31) | 10 (13) | 8 (12) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (4) | 6 (6) | 4 (5) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 8 (17) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 8 (9) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 16 (17) | 8 (11) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 14 (19) | 15 (23) | 7 (9) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 11 (13) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 22 (33) | 16 (30) | 5 (6) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 24 (33) | 12 (24) | 6 (6) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 22 (30) | 6 (9) | 2 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 7 (8) | 4 (5) | 2 (2) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 8 (8) | 3 (5) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 32 (65) | 2 (10) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (4) | 10 (29) | 2 (3) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 7 (7) | 17 (17) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 17 (48) | 2 (6) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 36 (49) | 57 (114) | 2 (2) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 11 (11) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (24) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 9 (18) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (25) | 23 (38) | 2 (4) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (11) | 6 (7) | 3 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (52) | 10 (11) | 12 (18) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (29) | 24 (27) | 11 (13) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 (9) | 5 (7) | 3 (3) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 12 (15) | 3 (7) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (21) | 11 (11) | 6 (7) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 24 (29) | 27 (54) | 6 (10) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 5 (5) | 13 (14) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 21 (26) | 22 (37) | 17 (27) | 0 (0) | 0 (0)
Hemiparaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 5 (7) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 28 (41) | 4 (4) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 6 (7) | 8 (10) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 31 (51) | 1 (1) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 9 (11) | 4 (6) | 4 (4) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Discouragement (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 12 (14) | 10 (11) | 7 (7) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (7) | 11 (28) | 2 (5) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (31) | 23 (26) | 7 (9) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (25) | 15 (22) | 6 (8) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 23 (30) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 8 (10) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 3 (3) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 6 (7) | 5 (6) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 13 (15) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 11 (11) | 29 (32) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (6) | 8 (22) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (21) | 14 (15) | 9 (11) | 3 (3) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 25 (35) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (37) | 12 (16) | 15 (24) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (12) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 19 (27) | 16 (22) | 10 (12) | 2 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (10) | 1 (2) | 0 (0) | 0 (0)
Superficial inflammatory dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 19 (25) | 16 (23) | 2 (2) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 3 (3) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT02563002/Prot_SAP_001.pdf